CLINICAL TRIAL: NCT06553092
Title: Turkish Validity and Reliability Study of Hospital for Special Surgery Shoulder Surgery Expectations Survey
Status: Not yet recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Principal Investigator, Gazi University
Other Study IDs: Iayas12
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Shoulder Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- urkish-Speaking Patients Undergoing Shoulder Surgery: This cohort consists of Turkish-speaking patients who have undergone shoulder surgery. Participants will complete the Turkish version of the Hospital for Special Surgery Shoulder Surgery Expectations Survey.
  Interventions: Other: Turkish Version of the Hospital for Special Surgery Shoulder Surgery Expectations Survey

INTERVENTIONS:
Other: Turkish Version of the Hospital for Special Surgery Shoulder Surgery Expectations Survey — The Hospital for Special Surgery (HSS) Shoulder Surgery Expectations Survey is a patient-reported outcome measure designed to assess a patient's expectations before undergoing shoulder surgery. It helps clinicians understand what patients anticipate regarding pain relief, functional improvement, and overall recovery from the procedure.The HSS Shoulder Surgery Expectations Survey contains 20 questions. Each question addresses a specific aspect of shoulder function or a potential outcome that patients might expect from their surgery.Each question is scored between 1-5.It is evaluated out of a total of 80 points. A higher score indicates a greater expectation of improvement.

SUMMARY:
This study aims to evaluate the Turkish validity and reliability of the Hospital for Special Surgery Shoulder Surgery Expectations Survey. By translating the original survey into Turkish and administering it to a sample of patients who have undergone shoulder surgery, the research seeks to determine whether the survey maintains its accuracy and consistency in the Turkish context. The study will involve statistical analyses to assess the survey's reliability, internal consistency, and construct validity, ensuring that the tool is culturally appropriate and effective for Turkish-speaking patients.

DETAILED DESCRIPTION:
The process begins with the translation of the original survey into Turkish, followed by a back-translation to ensure accuracy. The adapted survey is then reviewed by a panel of experts to confirm its cultural relevance and clarity.

Once finalized, the Turkish version of the survey is administered to a cohort of Turkish-speaking patients who have undergone shoulder surgery. Participants complete the survey at a designated time point, typically postoperatively, to assess their expectations and outcomes related to the surgery. The collected data are then analyzed to evaluate the survey's reliability (internal consistency, test-retest reliability) and validity (content, construct, and criterion validity) within this specific population.

The goal of the intervention is to ensure that the Turkish version of the survey is a reliable and valid tool for assessing patient expectations and satisfaction following shoulder surgery, making it suitable for use in clinical practice and research in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Underwent Shoulder Surgery
* Native Turkish Speakers
* Adults (18 years and older)
* Consent to Participate

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of native Turkish-speaking patients who have undergone shoulder surgery at various hospitals and clinics in Turkey. These patients will include adults of all ages, both male and female, who have received a diagnosis requiring surgical intervention for shoulder conditions such as rotator cuff tears, shoulder impingement, labral tears, or shoulder instability.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Validity and Reliability of the Turkish Version of the Hospital for Special Surgery Shoulder Surgery Expectations Survey | 6 months
  The primary outcome measure is to evaluate the psychometric properties of the Turkish version of the Hospital for Special Surgery Shoulder Surgery Expectations Survey. This includes assessing the survey's internal consistency, test-retest reliability, content validity, construct validity, and criterion validity in a cohort of Turkish-speaking patients who have undergone shoulder surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ulunay Kanatlı, Professor, Study Director — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No